CLINICAL TRIAL: NCT00633867
Title: Randomised Controlled Trial of Intubation With the McGrath Series 5 Video Laryngoscope vs the Macintosh Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Grampian (Other Government)
Responsible Party: Doctor William Brampton, NHS Grampian
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-so802-4
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2010-03-25 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2008-03

CONDITIONS: Tracheal Intubation
Keywords: Tracheal intubation; Laryngoscopy; videolaryngoscope; McGrath; success; time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation c McGrath videolaryngoscope (Active Comparator): Tracheal Intubation using McGrath video-laryngoscope
  Interventions: Device: McGrath
- Intubation using Macintosh Laryngoscope (Active Comparator): Tracheal intubation using Macintosh Laryngoscope
  Interventions: Device: Tracheal intubation using Macintosh Laryngoscope

INTERVENTIONS:
Device: McGrath — Tracheal intubation, using Mcgrath video-laryngoscope
  Other Names: Aircraft Medical McGrath Series 5 Video Laryngoscope
  Arms: Intubation c McGrath videolaryngoscope
Device: Tracheal intubation using Macintosh Laryngoscope — Tracheal intubation using Macintosh Laryngoscope
  Arms: Intubation using Macintosh Laryngoscope

SUMMARY:
The simplicity of use and intuitive function of the McGrath video-laryngoscope suggests it may have a bigger role than as a back-up to conventional direct laryngoscopy and could possibly be the first-line laryngoscope for situations where difficult intubations are more likely or more hazardous. The incidence of difficult or failed intubation for an individual anaesthetist is related to their experience, decreasing as experience increases. The purpose of this trial is to evaluate the McGrath laryngoscope when used by relatively inexperienced anaesthetists, who are those most likely to encounter difficulties.

The null hypotheses to be tested is that there is no difference between the Macintosh and McGrath laryngoscope in terms of ease and success in intubation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and over) scheduled for elective surgery whose anaesthetic plan would normally include oral intubation using a Macintosh laryngoscope blade after induction of general anaesthesia and who have given valid informed consent.

Exclusion Criteria:

* Patients requiring special techniques for intubation such as rapid sequence induction
* Adults who have learning difficulties
* Are unconscious or very severely ill
* Have a terminal illness; are in an emergency situation
* Have a mental illness
* Have dementia
* Prisoners
* Those who could be considered to have a particularly dependent relationship with the investigator and other vulnerable groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: william brampton, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Hospitals, NHS Grampian, Aberdeen, UK, United Kingdom

REFERENCES:
- [Result] Walker L, Brampton W, Halai M, Hoy C, Lee E, Scott I, McLernon DJ. Randomized controlled trial of intubation with the McGrath Series 5 videolaryngoscope by inexperienced anaesthetists. Br J Anaesth. 2009 Sep;103(3):440-5. doi: 10.1093/bja/aep191. Epub 2009 Jul 15. PMID 19605408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: adult patients undergoing elective tracheal intubation at induction of anaesthesia Between February and August 2008
Pre-assignment Details: 139 patients consented for study. 120 assigned to groups. 19 not studied: no McGrath® scope available (n=10). No direct supervision of intubator (n=6). Case cancellation or changes (n=3).
Groups:
- McGrath: Tracheal Intubation using McGrath video-laryngoscope
- Macintosh: Tracheal intubation using Macintosh Laryngoscope
Period: Overall Study
Arm/Group | McGrath | Macintosh
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | McGrath | Macintosh | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 48 [39 to 63.5] | 60.5 [41.3 to 70] | 54 [40 to 66.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  United Kingdom | 60 | 60 | 120

OUTCOME MEASURES:

1. Secondary Outcome: Difference in Learning to Use the Scopes
Description: Is there a difference between trainee anaesthetists in learning to use the scopes
Time Frame: At analysis
Reporting Status: Not Posted

2. Secondary Outcome: Quality of View of the Vocal Cords
Time Frame: At analysis
Reporting Status: Not Posted

3. Secondary Outcome: Number of Attempts to Secure Successful Intubation
Description: Is there a difference in the number of attempts required to secure successful intubation ?
Time Frame: At analysis
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Initial Oesophageal Intubation
Time Frame: At analysis
Reporting Status: Not Posted

5. Secondary Outcome: Number of Intubations Taking More Than 70 Seconds
Time Frame: At Analysis
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Low Arterial Saturation During Intubation
Time Frame: At analysis
Reporting Status: Not Posted

7. Secondary Outcome: Incidence of Visible Trauma to the Airway
Time Frame: At analysis
Reporting Status: Not Posted

8. Primary Outcome: Intubation Time
Description: Time from anaesthetist picking up laryngoscope until 1st upward capnograph deflection after intubation
Time Frame: At intubation
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | McGrath | Macintosh
Number analyzed (Participants) | 60 | 60
seconds | 47.0 [39.0 to 60.0] | 29.5 [23.0 to 36.8]
Statistical Analysis 1: Comparison: Macintosh; Test type: Superiority or Other; p < 0.01, Log Rank

ADVERSE EVENTS:
Arm/Group | McGrath | Macintosh
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No